CLINICAL TRIAL: NCT04526288
Title: A Randomized Trial for Patients With High-Grade Myeloid Neoplasms With Measurable Residual Disease (MRD): CPX-351 vs. Immediate Allogeneic Hematopoietic Cell Transplantation
Brief Title: CPX-351 Versus Immediate Stem Cell Transplantation for the Treatment of High-Grade Myeloid Cancers With Measurable Residual Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Filippo Milano, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1007476; NCI-2020-05619 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10545 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome With Excess Blasts-2; Myeloid Neoplasm
Keywords: Myeloid and Monocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Monocytic, Acute | interventions — Stem Cell Transplantation; CPX-351; Injections; Cytarabine; Daunorubicin; Liposomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (alloHCT) (Active Comparator): Patients undergo alloHCT.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation
- Arm B (CPX-351, alloHCT) (Experimental): Patients receive CPX-351 IV over 90 minutes on days 1, 3, and 5. Treatment may repeat for an additional cycle for a total of 2 cycles (on days 1 and 3 only of cycle 2) in the absence of disease progression or unacceptable toxicity. Within 60 days after completion of CPX-351, patients undergo alloHCT.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Liposome-encapsulated Daunorubicin-Cytarabine

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo alloHCT
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; Hematopoietic stem cell (HSC); Hematopoietic stem cell transplant (HSCT); Stem Cell Transplantation, Allogeneic
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal Cytarabine (AraC)-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos; Daunorubicin and Cytarabine (Liposomal)
  Arms: Arm B (CPX-351, alloHCT)

SUMMARY:
This phase II trial studies the effect of CPX-351 followed by donor stem cell transplantation versus immediate donor stem cell transplantation in treating patients with high-grade myeloid cancers with measurable residual disease. Chemotherapy drugs, such as CPX-351, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before donor stem cell transplantation may help kill cancer cells in the body and make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow.

DETAILED DESCRIPTION:
OUTLINE:

Patients are randomized to 1 of 2 arms.

Arm A: Patients undergo alloHCT.

Arm B: Patients receive CPX-351 intravenously (IV) over 90 minutes on days 1, 3, and 5. Treatment may repeat for an additional cycle for a total of 2 cycles (on days 1 and 3 only of cycle 2) in the absence of disease progression or unacceptable toxicity. Within 60 days after completion of CPX-351, patients undergo alloHCT.

After completion of study enrollment, patients will be followed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (AML) other than acute promyelocytic leukemia (APL), myelodysplastic syndrome with excess blasts-2 (MDS-EB2), or another high-risk myeloid neoplasm (>= 10% blasts in the blood or marrow), having completed at least one cycle of chemotherapy intended to induce remission
* Subjects must have MRD, defined as the presence of original disease detected by multi-parameter flow cytometry and cytogenetic/molecular assessment within 90 days of chemotherapy intended to induce remission:

  * Abnormal cells identified by multiparameter flow cytometry, present at a frequency of between 0% and 5% of total nucleated cells, judged in the opinion of the hematopathologist to represent continued presence of malignant cells
  * Abnormal karyotype; present in any number of metaphase cells
  * Abnormal fluorescence in-situ hybridization; judged in the opinion of the hematopathologist to represent continued presence of malignant cells
  * The presence of any leukemia associated mutation as detected by DNA sequencing, except mutations in DNMT3A, TET2 (tet methylcytosine dioxygenase 2), or ASXL1. This includes (but is not limited to) the following genes: CBL (CDS), CSF3R (colony stimulation factor 3 receptor; exons 14, 15, 17), EZH2 (exons 15-20), FBXW7 (CDS), FGFR1 (exons 4, 11-17, partial 18), FLT3 (FMS-like tyrosine kinase 3; p.D835H), GATA1 (exons 2-3), GATA2 (exons 3-5), HRAS (exon 1-2), IDH1 (isocitrate dehydrogenase NADP+ 1; p.R132), IDH2 (exon 4), JAK2 (Janus kinase 2; exon 12, 14, 16), KIT (8-18), KMT2A (CDS), KRAS (CDS), MAP2K1 (exons 2, 3, 6), MPL (exon 10), MYD88 (exon 3-5), NOTCH1 (exons 20, 26, 27), NPM1 (exon 12), NRAS (CDS), PDGFRA (exons 12-18), PHF6 (CDS), PTEN (CDS), RB1 (CDS), RUNX1 (exon 4-8), SF3B1 (exon 14-16), SRSF2 (exon 1), STAG2 (CDS), STAT3 (exons 20-21), TP53 (CDS), U2AF1 (exons 2, 6), WT1 (CDS), and ZRSR2 (CDS)
* Allowable prior therapy:

  * For the purposes of this study intensive chemotherapy will include regimens listed below. Additional regimens may be included at the discretion of the study principal investigator (PI)

    * Any regimen including cytarabine at a dose of 100 mg/m^2/day for at least 7 days and an anthracycline at any dose +/- gemtuzumab ozogamicin (GO)
    * Any regimen including cytarabine at a dose of at least 100 mg/m^2/day for at least 5 days and a purine analog at any dose (e.g. clofarabine, fludarabine, cladribine) +/- GO
* Ability to understand and voluntarily sign a written informed consent document (ICF)
* Absence of a concomitant illness with a likely survival of < 1 year
* Medically fit, defined as a treatment related mortality score (TRM) of =< 13.1 calculated according to Walter et al, Journal of Clinical Oncology (JCO) 2011
* Additionally, subjects should be eligible in the opinion of their treating physician for allogeneic transplantation
* Bilirubin =< 2.5 x institutional upper limit of normal, unless elevation is thought to be due to Gilberts syndrome or hemolysis (within 14 days of study start [unless otherwise noted] to be enrolled in the study)
* Left ventricular ejection fraction >= 40% assessed by multiple gated acquisition scan (MUGA), echocardiography or other appropriate diagnostic modality within 12 months of enrollment with no clinical evidence of decompensated congestive heart failure
* Creatinine clearance of >= 30 mL/min as measured by Cockcroft Gault equation (within 14 days of study start [unless otherwise noted] to be enrolled in the study)
* Consent of female patients with a negative serum or urine pregnancy test to use a medically acceptable method of contraception throughout the entire study period and for 6 months following the last dose of CPX-351
* Male patients must be willing to refrain from sperm donation for 6 months following the last dose of CPX-351 and must use adequate contraception throughout the entire study period and for 6 months following the last dose of CPX-351
* Patients enrolling in this trial should intend to complete the treatments described and should be eligible in the opinion of the treating physician for allogeneic transplantation
* Patients must have a caregiver capable of providing post-HCT care, who will be present once conditioning therapy begins
* The informed consent document (ICF) must be signed and dated by the subject or by the subject's legally authorized representative if the subject is unable to sign

Exclusion Criteria:

* Allogeneic myeloablative hematopoietic cell transplant within 6 months
* Autologous hematopoietic cell transplant within 6 months
* Known Hypersensitivity to CPX-351

  * Patients may not have known hypersensitivity to CPX-351, daunorubicin, cytarabine, or liposomal products
* Prior treatment with two or more cycles of CPX-351
* Treatment within the last 30 days of other investigational antineoplastic agents
* Evidence of organ dysfunction likely to preclude safe transplantation including the following:

  * Symptomatic coronary artery disease or uncontrolled arrhythmia within the prior 3 months and since most recent anthracycline exposure
  * Myocardial impairment of any cause resulting in heart failure as determined by New York (NY) Heart Association Criteria (class III or IV)
  * Corrected diffusion capacity of the lung for carbon monoxide (DLCOc) < 40% or forced expiratory volume in 1 second (FEV1) < 50%
  * Need for supplemental oxygen
* Active systemic fungal, bacterial, viral or other infection, unless under treatment with anti-microbials and/or controlled or stable (e.g. if specific, effective therapy is not available/feasible or desired [e.g. chronic viral hepatitis, human immunodeficiency virus (HIV)])
* Female patients who are pregnant, nursing, or lactating
* Patients with an inability to accept blood transfusions
* Inability to give informed consent, or unable to comply with the treatment protocol including appropriate supportive care, follow-up and tests
* Any other condition that would cause a risk to patients if they participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2023-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Milano, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients arrived to Fred Hutchinson Cancer Center, Transplant Clinic, for transplant screening and disease staging. Upon confirmation of ability to proceed to transplant and concurrent enrollment in transplant protocol, recruitment to this study was offered. The dates of the study's recruitment period were 3/16/2021-12/07/2022.
Groups:
- Arm A (alloHCT): Patients undergo allogeneic transplant (alloHCT) and do not receive investigational product.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo alloHCT
Period: Overall Study
Arm/Group | Arm A (alloHCT) | Arm B (CPX-351, alloHCT)
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Population: Single Arm A participant followed for survival only.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (alloHCT) | Arm B (CPX-351, alloHCT) | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The survival (in days) of subjects in the two arms will be compared using the log-rank test.
Time Frame: Up to 730 days post-randomization.
Population: We did not enroll sufficiently to allow for analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Arm A (alloHCT) | Arm B (CPX-351, alloHCT)
Number analyzed (Participants) | 1 | 0
Days | 730 (0) |

2. Secondary Outcome: Relapse-free Survival
Description: The following comparisons will be made: (1) number of days elapsing between the date of minimal residual disease (MRD) identification and the date of death or relapse, (2) among transplanted patients, the number of days elapsing between the date of transplantation and the date of death or relapse.
Time Frame: From the time of randomization up to 2 years post-randomization. For descriptive purposes, we shall also report survival and relapse-free survival from time of transplant up to 2 years post-transplant among patients who receive a transplant.
Population: Data was not collected for this outcome measure.
Arm/Group | Arm A (alloHCT) | Arm B (CPX-351, alloHCT)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Rate of Transplantation
Description: This outcome will be assessed among patients who have begun transplantation conditioning 60 days and 180 days following enrollment will be compared using the chi-squared test. The time to transplantation among the two arms will be compared by comparing the number of days elapsed between enrollment and the initiation of transplantation conditions by the log-rank test.
Time Frame: Up to 2 years post-randomization
Population: Data was not collected for this outcome measure because the one participant did not start transplantation conditioning.
Arm/Group | Arm A (alloHCT) | Arm B (CPX-351, alloHCT)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Frequencies of the Types of Transplantation Received
Description: Among the patients receiving transplantation, the proportion of patients in each arm receiving myeloablative transplantation conditioning will be compared using the chi-squared or Fisher's exact test. Among patients receiving transplantation, the proportion of patients in each arm receiving donor stem cells from a haploidentical donor, an unrelated donor, or from cord blood unit will each be compared using the chi-squared or Fisher's exact test.
Time Frame: Up to 2 years post-randomization
Population: The one participant enrolled did not proceed with transplant on the study.
Arm/Group | Arm A (alloHCT) | Arm B (CPX-351, alloHCT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) only collected for participants randomized to Arm B of the study and receiving the investigational agent (CPX-351). Adverse events will be tracked for up to 56 days after the last dose of CPX-351 or until resolution. Collection of AEs should cease with the start of any new therapy or conditioning for transplant.
Description: Events not considered AEs in this study:
  * Disease progression or relapse
  * Medical conditions present at screening
  * Abnormal laboratory values outside of normal laboratory parameters
  * Diagnostic tests and medical or surgical procedures
  * Preplanned hospitalizations
Arm/Group | Arm A (alloHCT) | Arm B (CPX-351, alloHCT)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Low accrual lead to early termination of the study. The single individual enrolled was randomized to the non-investigational arm of the study (Arm A) and was removed from the study prior to conditioning which only allowed for follow-up of overall survival. Therefore, there is little to no interpretable data to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT04526288/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT04526288/ICF_000.pdf